CLINICAL TRIAL: NCT02965105
Title: Clinical Study Investigating Safety and Performance of a New Urinary Intermittent Catheters in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CP271
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Incontinence, Urinary
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast Test Catheter; then Speedicath (Experimental): The subjects allocated to this arm first test Coloplast Test Catheter and then after cross over test the comparator Speedicath Catheter
  Interventions: Device: Coloplast Test Catheter; Device: Speedicath
- First Speedicath; then Coloplast Test Catheter (Experimental): The subjects allocated to this arm first test Speedicath Catheter and then after cross over test Coloplast Test Catheter
  Interventions: Device: Coloplast Test Catheter; Device: Speedicath

INTERVENTIONS:
Device: Coloplast Test Catheter — This is a newly developed intermittent catheter
Device: Speedicath — This is a marketed Catheter which is used as comparator

SUMMARY:
The aim of the study is to test the performance and safety of a newly developed intermittent catheter

ELIGIBILITY:
Inclusion Criteria:

* 1. Have given written informed consent and signed letter of authority 2. Be at least 18 years of age and have full legal capacity 3. Be a male 4. Willing to refrain from using analgetics up to 24 hours prior to catheterization visits 5. Have a negative urine multistix - erythrocytes (Microscopic haematuria) 6. Have a negative urine multistix:

  * Leukocytes
  * Nitrite Or if positive, subsequent negative for bacterial growth in urine culture

Exclusion Criteria:

1. Abnormalities, diseases or surgical procedures performed in the lower urinary tract
2. Symptoms of urinary tract infections (at least one of the following: frequent urination, stinging or pain at urination)
3. Participating in other clinical investigations related to urinary tracts system during this investigation (inclusion to termination) or have previously participated in this investigation
4. Known hypersensitivity toward any of the test products -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain | 1 day
  Pain experienced by the subjects at catheterisation is measure with the VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — MD at the clinic for urology at Rigshospitalet
Locations (1):
- Rigshopsitalet, Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No